CLINICAL TRIAL: NCT02579343
Title: Adjunctive Treatment of Major Depression Utilizing Auricular Acupuncture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Florida Gulf Coast University (Other)
Responsible Party: Principal Investigator, Sherry Alexander, Research Compliance Coordinator, Florida Gulf Coast University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FloridaGCU
Record Dates: First submitted 2015-10-05; First posted 2015-10-19 (Estimated); Results first posted 2021-10-12 (Actual); Last update posted 2021-10-12 (Actual); Status verified 2021-09

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Acupuncture, Ear; Escitalopram

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Auricular Acupuncture + Lexapro (Experimental): Participants will be treated with the SSRI Lexapro 10 mg daily which will be increased to 20 mg daily at week 2. Participants in this group will be treated twice weekly during their follow-up visits with micro-currents of electricity through auricular acupuncture.
  Interventions: Device: Auricular Acupuncture
- Sham Auricular Acupuncture + Lexapro (Sham Comparator): Participants will be treated with the SSRI Lexapro 10 mg daily which will be increased to 20 mg daily at week 2. Participants will be treated twice weekly during their follow-up visits with sham auricular acupuncture (No micro-current).
  Interventions: Drug: Sham Auricular Acupuncture + Lexapro

INTERVENTIONS:
Device: Auricular Acupuncture — Auricular acupuncture is a form of acupuncture which utilizes the surface of the external ear to identify points of inflammation in the body. It does this, in this case, by utilizing the Pointer Excel II probe which can pick up a change in electrical conductivity on the surface of the ear, which reflects an internal point of inflammation or stress. Once the point of inflammation is identified, the Pointer Excel II is equipped with a sensor that it will not only illuminate by way of a small light on the front of the probe will also identify the point of inflammation by way of an auditory signal. Once the point of inflammation is identified auricular acupuncture will treat that point with a micro-current of electricity for several seconds.
  Other Names: Pointer Excel II
  Arms: Auricular Acupuncture + Lexapro
Drug: Sham Auricular Acupuncture + Lexapro — Participants will be treated with the SSRI Lexapro 10 mg daily which will be increased to 20 mg daily at week 2. Participants will be treated twice weekly during their follow-up visits with sham auricular acupuncture (No micro-current).
  Other Names: SSRI Lexapro
  Arms: Sham Auricular Acupuncture + Lexapro

SUMMARY:
This will be a randomized, single blind study of 6 weeks duration involving the use of auricular acupuncture or sham acupuncture in the adjunctive treatment of depression in college students.

DETAILED DESCRIPTION:
This will be a randomized, single blind study of 6 weeks duration involving the use of auricular acupuncture or sham acupuncture in the add adjunctive treatment of depression in college students. College students presenting for care at Counseling and Psychological Services, who meet Diagnostic and Statistical Manual of Mental Disorders - V (DSM-V) criteria for major depression single episode or recurrent will be included in the trial. Subjects will be randomized into a sham auricular acupuncture group, or a treatment acupuncture group. All subjects who meet the inclusion criteria will be treated with the Selective serotonin reuptake inhibitor (SSRI) Lexapro 10 mg daily which will be increased to 20 mg daily at week 2. Some subjects will be treated twice weekly during their follow-up visits with sham auricular acupuncture, some subjects will be treated with micro-currents of electricity in the auricular acupuncture group. The duration of the trial will be 6 weeks.

Auricular acupuncture is a form of acupuncture which utilizes the surface of the external ear to identify points of inflammation in the body. It does this, in this case, by utilizing the Pointer Excel II probe which can pick up a change in electrical conductivity on the surface of the ear, which reflects an internal point of inflammation or stress. Once the point of inflammation is identified, the Pointer Excel II is equipped with a sensor that it will not only illuminate by way of a small light on the front of the probe will also identify the point of inflammation by way of an auditory signal. Once the point of inflammation is identified auricular acupuncture will treat that point with a micro-current of electricity for several seconds. In the case of treatment, there will be an auditory alarm followed by a micro -current dose of electricity. Sham acupuncture will be characterized by the auditory alarm, but no current will be applied to the participants ear.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-V criteria for major depression single episode or recurrent as a primary diagnosis. Participants must have been symptomatic with depression for 2 months or more and less than 18 months.

Exclusion Criteria:

* a current diagnosis or history of alcohol or substance abuse or dependence that has not been in full and sustained remission for 3 months
* any current psychiatric diagnosis which is the primary focus of treatment other than major depression
* current history of mania or hypomania, schizophrenia, or any psychotic disorder, obsessive-compulsive disorder, autism spectrum conditions, organic mental disorders or mental disorders due to a physical condition
* the participant has a history of lack of response to a previous adequate treatment with 2 antidepressants for major depression at a standard dose for at least a six-week period of time
* any axis II disorder
* if the participant is female the participant agrees to use adequate contraception from the signing of the informed consent and throughout the study and for 30 days afterwards. pregnant or lactating females or those intending to become pregnant during the study are excluded
* if the participant is unlikely to comply with a clinical study protocol or is unsuitable for the study as determined by the principal investigator
* if the participant has clinically significant unstable physical illness such as neurologic disorders, diabetes, immunologic disorders, or any disturbance of a metabolic nature which may compromise the study
* the participant has a risk of suicide according to the investigators clinical judgment and according to the screening instruments used in the trial
* the subject has started receiving formal cognitive psychotherapy within 30 days from screening or plans to initiate such therapy during the study.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2015-08; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Prater, DO, Principal Investigator — Counseling and Psychological Services
Locations (1):
- Counseling and Psychological Services, Fort Myers, Florida, United States

REFERENCES:
- [Background] Berman BM, Lao L, Langenberg P, Lee WL, Gilpin AM, Hochberg MC. Effectiveness of acupuncture as adjunctive therapy in osteoarthritis of the knee: a randomized, controlled trial. Ann Intern Med. 2004 Dec 21;141(12):901-10. doi: 10.7326/0003-4819-141-12-200412210-00006. PMID 15611487
- [Background] Gori L, Firenzuoli F. Ear acupuncture in European traditional medicine. Evid Based Complement Alternat Med. 2007 Sep;4(Suppl 1):13-6. doi: 10.1093/ecam/nem106. PMID 18227925
- [Background] MacPherson H, Richmond S, Bland M, Brealey S, Gabe R, Hopton A, Keding A, Lansdown H, Perren S, Sculpher M, Spackman E, Torgerson D, Watt I. Acupuncture and counselling for depression in primary care: a randomised controlled trial. PLoS Med. 2013;10(9):e1001518. doi: 10.1371/journal.pmed.1001518. Epub 2013 Sep 24. PMID 24086114
- [Background] Nixon MK, Cheng M, Cloutier P. An open trial of auricular acupuncture for the treatment of repetitive self-injury in depressed adolescents. Can Child Adolesc Psychiatr Rev. 2003 Feb;12(1):10-2. PMID 19030475
- [Background] Qu SS, Huang Y, Zhang ZJ, Chen JQ, Lin RY, Wang CQ, Li GL, Wong HK, Zhao CH, Pan JY, Guo SC, Zhang YC. A 6-week randomized controlled trial with 4-week follow-up of acupuncture combined with paroxetine in patients with major depressive disorder. J Psychiatr Res. 2013 Jun;47(6):726-32. doi: 10.1016/j.jpsychires.2013.02.004. Epub 2013 Mar 14. PMID 23498306
- [Background] Sinyor M, Schaffer A, Levitt A. The sequenced treatment alternatives to relieve depression (STAR*D) trial: a review. Can J Psychiatry. 2010 Mar;55(3):126-35. doi: 10.1177/070674371005500303. PMID 20370962
- [Background] Wang SM, Peloquin C, Kain ZN. The use of auricular acupuncture to reduce preoperative anxiety. Anesth Analg. 2001 Nov;93(5):1178-80, table of contents. doi: 10.1097/00000539-200111000-00024. PMID 11682391

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period began during the summer of 2015 and continued through the spring of 2016. All participants were recruited through Counseling and Psychological Services.
Pre-assignment Details: Two potential participants immediately dropped from study prior to group assignment related to scheduling and commitment concerns.
Groups:
- Auricular Acupuncture + Lexapro: Participants will be treated with the SSRI Lexapro 10 mg daily which will be increased to 20 mg daily at week 2. Participants in this group will be treated twice weekly during their follow-up visits with micro-currents of electricity through auricular acupuncture.
  Auricular Acupuncture: Auricular acupuncture is a form of acupuncture which utilizes the surface ear to identify points of inflammation in the body. It does this by utilizing the Pointer Excel II probe which can pick up a change in electrical conductivity on the surface of the ear, which reflects an internal point of inflammation. Once the point of inflammation is identified, the Pointer Excel II is equipped with a sensor that it will not only illuminate by way of a small light on the front of the probe will also identify the point of inflammation by way of an auditory signal. Once the point of inflammation is identified auricular acupuncture will treat that point with a micro-current of electricity for several seconds.
Period: Overall Study
Arm/Group | Auricular Acupuncture + Lexapro | Sham Auricular Acupuncture + Lexapro
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Auricular Acupuncture + Lexipro: Participants will be treated with the SSRI Lexapro 10 mg daily which will be increased to 20 mg daily at week 2. Participants in this group will be treated twice weekly during their follow-up visits with micro-currents of electricity through auricular acupuncture.
  Auricular Acupuncture: Auricular acupuncture is a form of acupuncture which utilizes the surface ear to identify points of inflammation in the body. It does this by utilizing the Pointer Excel II probe which can pick up a change in electrical conductivity on the surface of the ear, which reflects an internal point of inflammation. Once the point of inflammation is identified, the Pointer Excel II is equipped with a sensor that it will not only illuminate by way of a small light on the front of the probe will also identify the point of inflammation by way of an auditory signal. Once the point of inflammation is identified auricular acupuncture will treat that point with a micro-current of electricity for several seconds.
- Total: Total of all reporting groups
Arm/Group | Auricular Acupuncture + Lexipro | Sham Auricular Acupuncture + Lexapro | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 1 | 8
  Male | 0 | 5 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 4 | 4 | 8
  Unknown or Not Reported | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 0 | 0 | 0
  White | 5 | 4 | 9
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Score of the Sheehan Disability Scale Through 6 Weeks
Description: Instrument developed to assess functional impairment in three inter-related domains; work/school, social and family life. Items are scored on a 0 - 10 point scale. Higher scores indicate more functional impairment.
Time Frame: Assessed at baseline and 6 weeks.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupuncture + Lexipro | Sham Auricular Acupuncture + Lexapro
Number analyzed (Participants) | 7 | 6
units on a scale
  Work / School Domain | -3.57 (1.03) | -1.5 (1.19)
  Social Life Domain | -2.29 (1.16) | -1.0 (1.20)
  Family Life Domain | -3.42 (1.14) | -0.17 (0.70)
Statistical Analysis 1: Comparison: Auricular Acupuncture + Lexipro vs Sham Auricular Acupuncture + Lexapro; Test type: Superiority; p = .05, Repeated Measures Analysis of Variance — P-value above was calculated. Does not reference threshold for clinical significance

2. Primary Outcome: Change of Mean Score of the Behavioral Health Measure-20 Between Baseline and End of Study
Description: The Behavioral Health Measure - 20 (BHM-20) is a 20-item client-report questionnaire that assesses the three phases of behavioral health: (a) well-being (distress, life satisfaction, motivation), (b) psychological symptoms (depression, anxiety, panic disorder, mood swings associated with bipolar disorder, eating disorder, alcohol/drug abuse, suicidality, risk of violence), and (c) life functioning (work/school, intimate relationships, social relationships, life enjoyment). The BHM-20 assesses the most frequently seen problems in outpatient psychotherapy. Scores range from 0-4. Lower scores indicate more distress.
Time Frame: Assessed at Baseline and After Treatment, Approximately 6 Weeks later.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Auricular Acupuncture + Lexipro | Sham Auricular Acupuncture + Lexapro
Number analyzed (Participants) | 7 | 6
units on a scale | 0.89 (0.280) | 0.47 (0.348)
Statistical Analysis 1: Comparison: Auricular Acupuncture + Lexipro vs Sham Auricular Acupuncture + Lexapro; Test type: Superiority; p = .05, Repeated Measures Analysis of Variance

ADVERSE EVENTS:
Time Frame: Adverse events were assessed throughout the duration of data collection for each individual (up to 6 weeks from baseline, initial assessment).
Arm/Group | Auricular Acupuncture + Lexipro | Sham Auricular Acupuncture + Lexapro
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

LIMITATIONS AND CAVEATS:
Main limitation related to small sample size due to difficulties with recruitment. Please interpret results with care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes